CLINICAL TRIAL: NCT05705895
Title: Evaluation of the Efficiency of the Central Venous Catheter Care Protocol for Patients With Hematopoietic Stem Cell Transplantation
Brief Title: The Efficiency of the Central Venous Catheter Care Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Canan Yaranoglu, Nurse, MsN, RN, Principle Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/51
Record Dates: First submitted 2023-01-13; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Stem Cell Transplant Complications; Central Venous Catheter Exit Site Infection
Keywords: Central Venous Catheter; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients and care providers know which group they are in, but the outcome assessor does not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Catheter care is provided in line with the CVC care protocol developed by the researcher.
  Interventions: Procedure: CENTRAL VENOUS CATHETER CARE PROTOCOL
- Control Group (No Intervention): No intervention will be made to the patients in the control group, and catheter care will be provided in line with the clinical routine.

INTERVENTIONS:
Procedure: CENTRAL VENOUS CATHETER CARE PROTOCOL — Catheter care is provided in line with the CVC care protocol developed by the researcher:
  * For subsequent catheter care, a transparent sterile catheter cover impregnated with 2% chlorhexidine gluconate will be used.
  * The entry point of the catheter will be wiped with a disposable sterile skin cleaning applicator containing 2% Chlorhexidine Gluconate and 70% Isopropyl Alcohol, which will be provided by the researchers, and wait for it to dry.
  * Vein valve/needleless connector will be used.
  * Effective manual disinfection of needle-free connectors (hubs) will be ensured before each intervention.
  * Needle-free connectors will be replaced every 96 hours at the latest.
  * If necessary, the catheter lumen will be washed with a disposable, positive-pressure sterile washing system containing 10 ccs 0.9% sodium chloride to be provided by the investigators.
  * Pulsatile "give stop give stop" technique will be used in the washing process.
  Arms: Intervention Group

SUMMARY:
The study aims to evaluate the effectiveness of a central venous catheter (CVC) care protocol, which was created using current guidelines, research results, and expert opinions, on developing CVC-related bloodstream infection in patients with hematopoietic stem cell transplantation (HSCT) until discharge.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is one of the important treatment approaches that prolongs survival in patients with hematological malignancies, immunodeficiency and some solid tumors. Despite advances in the treatment process, reasons such as recurrence of the underlying disease, organ toxicities and infectious complications adversely affect treatment success. Reasons such as high-dose chemotherapy, frequent blood sampling, stem cell reinfusion, and total parenteral nutrition applied to HSCT patients increase the need for central venous catheter insertion. Although these tools are often necessary and useful in the bone marrow transplantation process, they also bring mechanical, embolic, and infectious complications.

Central venous catheters (CVC) are one of the main applications of modern clinical treatment. Reasons such as high-dose chemotherapy, frequent blood sampling, stem cell reinfusion, and total parenteral nutrition applied to HSCT patients increase the need for central venous catheter insertion. Although these tools are often necessary and valuable in the bone marrow transplantation process, they also bring mechanical, embolic, and infectious complications. The study aims to evaluate the effectiveness of a central venous catheter (CVC) care protocol, created using current guidelines, research results, and expert opinions, on developing CVC-related bloodstream infection in patients with hematopoietic stem cell transplantation (HSCT) until discharge.

This research is a pretest-posttest quasi-experimental clinical study. It is conducted with 60 patients between January 2022 and December 2023. The data is collected with Patient Information Form and Daily Patient Evaluation Chart. No application will be made to 30 patients in the control group, and catheter care will be provided to the patients of the intervention group in line with the CVC Care Protocol created by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized by the Medical Oncology Clinic at in a training and research hospital to become an Autologous HSCT,
* The patient has an 8F-size, two-lumen temporary CVC,
* Over 18 years of age
* There is no communication problem,
* Agreeing to participate in the research voluntarily after being informed about the study,

Exclusion Criteria:

* Using a vascular access method other than an 8F size two-lumen temporary CVC in the patient,
* Refusal to participate in the research voluntarily after being informed about the study,
* Identification of a different focus of infection in the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Descriptive Information Form | Baseline
  It was developed by the researchers by examining the literature; It contains information about the socio-demographic characteristics of the patients such as age, gender, marital status, educational status, and the planned chemotherapy protocol, previous treatments, and medical conditions such as chronic diseases. There are 8 questions in the first part of the form, which includes socio-demographic characteristics, and 12 questions in the second part, which includes information on medical status..
Daily Patient Evaluation Chart | During the procedure
  It was developed by researchers by examining the literature; patients' vital signs (recording of signs of infection such as hypotension, tachycardia, high fever), height-weight measurement results, daily central venous catheter insertion site control results (evaluation findings such as exudate, swelling, redness, discharge, etc.) and routine clinical procedures from patients every day. This is the chart in which the results of whole blood, CRP, Procalcitonin, sedimentation count values and hemoculture routinely taken at every fever, urine culture and catheter tip culture taken during discharge will be recorded. It also includes the control of the protocol implementation steps.

CONTACTS AND LOCATIONS:
Overall Officials: Canan PORUCU, MsN, RN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Science University Gülhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callister D, Limchaiyawat P, Eells SJ, Miller LG. Risk factors for central line-associated bloodstream infections in the era of prevention bundles. Infect Control Hosp Epidemiol. 2015 Feb;36(2):214-6. doi: 10.1017/ice.2014.32. PMID 25633005
- [Background] Demiraslan H, Cevahir F, Berk E, Metan G, Cetin M, Alp E. Is surveillance for colonization of carbapenem-resistant gram-negative bacteria important in adult bone marrow transplantation units? Am J Infect Control. 2017 Jul 1;45(7):735-739. doi: 10.1016/j.ajic.2017.01.006. Epub 2017 Feb 15. PMID 28214159
- [Background] Ferroni A, Gaudin F, Guiffant G, Flaud P, Durussel JJ, Descamps P, Berche P, Nassif X, Merckx J. Pulsative flushing as a strategy to prevent bacterial colonization of vascular access devices. Med Devices (Auckl). 2014 Nov 7;7:379-83. doi: 10.2147/MDER.S71217. eCollection 2014. PMID 25404862
- [Background] Gunasegaran N, See MTA, Leong ST, Yuan LX, Ang SY. A Randomized Controlled Study to Evaluate the Effectiveness of 2 Treatment Methods in Reducing Incidence of Short Peripheral Catheter-Related Phlebitis. J Infus Nurs. 2018 Mar/Apr;41(2):131-137. doi: 10.1097/NAN.0000000000000271. PMID 29489709
- [Background] Flint AC, Toossi S, Chan SL, Rao VA, Sheridan W. A Simple Infection Control Protocol Durably Reduces External Ventricular Drain Infections to Near-Zero Levels. World Neurosurg. 2017 Mar;99:518-523. doi: 10.1016/j.wneu.2016.12.042. Epub 2016 Dec 22. PMID 28012890